CLINICAL TRIAL: NCT06047080
Title: A Phase III, Multicenter, Randomized, Open-Label Study Comparing the Efficacy and Safety of Glofitamab (RO7082859) in Combination With Polatuzumab Vedotin Plus Rituximab, Cyclophosphamide, Doxorubicin, and Prednisone (Pola-R-CHP) Versus Pola-R-CHP in Previously Untreated Patients With Large B-Cell Lymphoma
Brief Title: An Open-Label Study Comparing Glofitamab and Polatuzumab Vedotin + Rituximab, Cyclophosphamide, Doxorubicin, and Prednisone Versus Pola-R-CHP in Previously Untreated Patients With Large B-Cell Lymphoma
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GO44145
Record Dates: First submitted 2023-09-14; First posted 2023-09-21 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Large B-Cell Lymphoma
MeSH Terms: interventions — glofitamab; polatuzumab vedotin; Rituximab; Cyclophosphamide; Doxorubicin; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Glofitamab + Pola-R-CHP (Experimental): Participants will receive glofitamab in combination with polatuzumab vedotin, rituximab, cyclophosphamide, doxorubicin, and prednisone (Pola-R-CHP).
  Interventions: Drug: Glofitamab; Drug: Polatuzumab vedotin; Drug: Rituximab; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Prednisone
- Pola-R-CHP (Active Comparator): Participants will receive Pola-R-CHP.
  Interventions: Drug: Polatuzumab vedotin; Drug: Rituximab; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Prednisone

INTERVENTIONS:
Drug: Glofitamab — Participants will receive intravenous (IV) glofitamab
  Arms: Glofitamab + Pola-R-CHP
Drug: Polatuzumab vedotin — Participants will receive IV polatuzumab vedotin in combination with R-CHP
Drug: Rituximab — Participants will receive IV rituximab
Drug: Cyclophosphamide — Participants will receive cyclophosphamide as part of CHP chemotherapy
Drug: Doxorubicin — Participants will receive IV doxorubicin
Drug: Prednisone — Participants will receive oral prednisone as part of CHP chemotherapy

SUMMARY:
The purpose of this study is to compare the efficacy and safety of glofitamab in combination with polatuzumab vedotin plus rituximab, cyclophosphamide, doxorubicin, and prednisone (Pola-R-CHP) vs Pola-R-CHP in participants with previously untreated CD20-positive large B-cell lymphoma (LBCL).

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated participants with CD20-positive LBCL
* Ability to provide tumor tissue
* International prognostic index (IPI) score 2-5
* Eastern cooperative oncology group (ECOG) performance status of 0, 1, or 2
* At least one bi-dimensionally measurable lesion, defined as > 1.5 cm in its longest dimension as measured by CT or MRI
* Left ventricular ejection fraction (LVEF) >/=50% on cardiac multiple-gated acquisition (MUGA) scan or cardiac echocardiogram (ECHO)
* Adequate hematologic function
* Negative HIV test at screening with exceptions as defined by the protocol
* Negative SARS-CoV-2 antigen or PCR test

Exclusion Criteria:

* Contraindication to any of the individual components of Pola-R-CHP or glofitamab, including prior receipt of anthracyclines, or history of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies, or known sensitivity or allergy to murine products
* Prior solid organ transplantation
* Participants receiving systemic immunosuppressive agent such as, but not limited to cyclosporin, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor agents within 4 weeks prior to first dose of study treatment
* Current Grade > 1 peripheral neuropathy by clinical examination or demyelinating form of Charcot-Marie-Tooth disease
* History of indolent lymphoma (e.g., Follicular Lymphoma, Marginal Zone Lymphoma, Waldenstrom macroglobulinemia)
* Current diagnosis of the following: Follicular lymphoma grade 3B; transformations of indolent B-cell lymphomas (e.g., de novo transformed follicular lymphoma); mediastinal grey zone lymphoma; primary mediastinal (thymic) large B-cell lymphoma; Burkitt lymphoma; primary large B-cell lymphoma of immune-privileged sites (encompassing primary diffuse large B-cell lymphoma of the CNS, primary large B-cell lymphoma of the vitreoretina and primary large B-cell lymphoma of the testis); primary effusion DLBCL; and primary cutaneous DLBCL, leg type
* Primary or secondary CNS lymphoma at the time of recruitment or history of CNS lymphoma
* Prior treatment with systemic immunotherapeutic agents
* Prior use of any monoclonal antibody for the purposes of treating cancer within 3 months of the start of Cycle 1
* Any investigational therapy for the purposes of treating cancer within 28 days prior to the start of Cycle 1
* Prior radiotherapy to the mediastinal/pericardial region
* Prior therapy for LBCL, with the exception of corticosteriods
* Corticosteroid use > 30 mg/day of prednisone or equivalent, for purposes other than lymphoma symptom control
* History of other malignant or non-malignant diseases that could affect compliance with the protocol or interpretation of results
* Significant or extensive history of cardiovascular disease
* Recent major surgery (within 4 weeks prior to the start of Cycle 1), other than for diagnosis
* Current or past history of central nervous system (CNS) disease, such as stroke, epilepsy, CNS vasculitis, or neurodegenerative disease
* Known or suspected chronic active Epstein-Barr viral infection
* Known or suspected history of hemophagocytic lymphohistiocytosis (HLH)
* Active autoimmune disease requiring treatment
* Clinically significant liver disease
* Live, attenuated vaccine within 4 weeks before study treatment infusion on Day 1 of Cycle 1 or anticipation that such a live, attenuated vaccine will be required during the study. Live vaccines during the study and until participants B cells recover are prohibited
* Any active infection within 7 days prior to Cycle 1 Day 1 that would impact participant safety
* Suspected active or latent tuberculosis
* Positive test results for chronic hepatitis B infection, hepatitis C, or the human T-lymphotropic virus type 1 (HTLV-1)
* History of progressive multifocal leukoencephalopathy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1130 (Actual)
Dates: Start 2023-09-18 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) as determined by Independent Review Facility (IRF) | From randomization to the first occurrence of disease progression or relapse, or death due to any cause, whichever occurs first (up to approximately 65 months)

SECONDARY OUTCOMES:
PFS as determined by the investigator | From randomization to the first occurrence of disease progression or relapse or death from any cause, whichever occurs first (up to approximately 65 months)
PFS as determined by the investigator and IRF for participants with international prognostic index (IPI) 3-5 | From randomization to the first occurrence of disease progression or relapse or death from any cause, whichever occurs first (up to 65 months)
Event-free survival efficacy causes (EFSeff) | From randomization to the earliest occurrence of disease progression or relapse; death due to any cause; initiation of new anti-lymphoma treatment; or positive biopsy for residual disease after treatment completion (up to approximately 65 months)
Complete response (CR) rate | At the end of treatment (up to approximately 65 months)
Objective response rate (ORR) | At treatment completion or discontinuation (up to approximately 65 months)
Overall survival (OS) | From randomization to death from any cause (up to approximately 65 months)
Duration of response (DOR) | From the first occurrence of a documented objective response to disease progression or death from any cause, whichever occurs first (up to approximately 65 months)
Duration of complete response (DOCR) | From the first occurrence of a documented complete response (CR) to disease progression or death, whichever occurs first (up to approximately 65 months)
Disease-free survival (DFS) | From a documented CR at the end of treatment to disease progression or death, whichever occurs first (up to approximately 65 months)
Serum concentration of glofitamab | Up to approximately 65 months
Incidence of anti-drug antibodies (ADAs) | Baseline up to approximately 65 months
Proportion of participants experiencing a clinically meaningful improvement in physical functioning and fatigue (EORTC QLQ-C30) and lymphoma symptoms (FACT-Lym LymS) | Up to approximately 65 months
Time to deterioration in physical functioning and fatigue (EORTC QLQ-C30) and lymphoma symptoms (FACT-Lym LymS) | Up to approximately 65 months
Percentage of Participants with Adverse Events (AEs) | From randomization to the end of study (up to approximately 65 months)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (231):
- United States (60):
  - Alaska Oncology & Hematology, LLC, Anchorage, Alaska
  - Kaiser Permanente - Anaheim (E. La Palma), Anaheim, California
  - University of California, San Francisco-Fresno, Clovis, California
  - City of Hope National Medical Center, Duarte, California
  - City of Hope - Lennar Foundation Cancer Center, Irvine, California
  - Valkyrie Clinical Trials, Los Angeles, California
  - UCLA Jonsson Comprehensive Cancer Center, Los Angeles, California
  - Kaiser Permanente - Roseville, Roseville, California
  - Kaiser Permanente - Santa Clara, Santa Clara, California
  - Stanford Univ School of Med, Stanford, California
  - Kaiser Permanente Medical Ctr, Vallejo, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - Rocky Mountain Cancer Center - Denver, Littleton, Colorado
  - Yale University School Of Medicine, New Haven, Connecticut
  - Medstar Franklin Square Medical Center, Washington D.C., District of Columbia
  - Miami Cancer Institute of Baptist Health, Inc., Miami, Florida
  - Memorial Cancer Institute at Memorial West, Pembroke Pines, Florida
  - Hawaii Cancer Care, Honolulu, Hawaii
  - Robert H. Lurie Comprehensive Cancer Center of Northwestern University, Chicago, Illinois
  - Illinois Cancer Care, Peoria, Illinois
  - Springfield Clinic, Springfield, Illinois
  - University of Iowa, Iowa City, Iowa
  - Ascension Via Christi Research, Wichita, Kansas
  - Ochsner Medical Center, New Orleans, Louisiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Henry Ford Health System, Novi, Michigan
  - M Health Fairview University of Minnesota Medical Center, Minneapolis, Minnesota
  - St. Luke's Hospital, Chesterfield, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - NYU Langone Hospital?Brooklyn, Brooklyn, New York
  - NYU Long Island Hospital, Mineola, New York
  - New York University Medical Center PRIME, New York, New York
  - Memorial Sloan Kettering Cancer Center David H Koch Center for Cancer Care, New York, New York
  - Weill Cornell Medical College-New York Presbyterian Hospital, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - North Shore Hematology Oncology Association PC, Shirley, New York
  - Montefiore Medical Center, The Bronx, New York
  - New York Cancer & Blood Specialists, The Bronx, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Levine Cancer Institute, Charlotte, North Carolina
  - Willamette Valley Cancer Insitute and Research Center, Springfield, Oregon
  - Kimmel Cancer Center Thomas Jefferson University, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - West Penn Hospital, Pittsburgh, Pennsylvania
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Greco-Hainesworth Tennessee Oncology Centers for Research, Chattanooga, Tennessee
  - West Cancer Center & Research Institute, Germantown, Tennessee
  - Tennessee Oncology, Nashville, Tennessee
  - Texas Oncology - Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - USOR - Texas Oncology - San Antonio Northeast, San Antonio, Texas
  - University of Vermont, Burlington, Vermont
  - Virginia Cancer Specialists, Fairfax, Virginia
  - Virginia Oncology Associates, Newport News, Virginia
  - Swedish Medical Center, Seattle, Washington
  - University of Washington - Seattle Cancer Care Alliance, Seattle, Washington
  - West Virginia University, Morgantown, West Virginia
  - Univ of Wisconsin Hosp & Clin, Madison, Wisconsin
- Argentina (4):
  - Instituto Alexander Fleming, Buenos Aires
  - FUNDALEU, Buenos Aires
  - Hospital Aleman de Buenos Aires, Buenos Aires
  - Sanatorio Allende, Córdoba
- Australia (11):
  - Concord Repatriation General Hospital, Concord, New South Wales
  - Prince of Wales Hospital- Department of Hematology, Randwick, New South Wales
  - Townsville Hospital, Douglas, Queensland
  - Princess Alexandra Hospital Woolloongabba, Woolloongabba, Queensland
  - Flinders Medical Centre, Bedford Park, South Australia
  - Royal Hobart Hospital, Hobart, Tasmania
  - Eastern Health, Box Hill, Victoria
  - St Vincent's Hospital Melbourne, Fitzroy, Victoria
  - Barwon Health, Geelong, Victoria
  - Peter Maccallum Cancer Centre, Melbourne, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
- Belgium (4):
  - Institut Jules Bordet, Anderlecht
  - UZ Brussel, Brussels
  - AZ Groeninge, Kortrijk
  - CHU de Liège (Sart Tilman), Liège
- Brazil (3):
  - Hospital Erasto Gaertner, Curitiba, Paraná
  - Instituto D'Or Pesquisa e Ensino, São Paulo, São Paulo
  - Hospital das Clinicas - FMUSP, Oncologia, São Paulo, São Paulo
- Canada (5):
  - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - William Osler Health Centre - Brampton Civic Hospital, Brampton, Ontario
  - Health Sciences North, Greater Sudbury, Ontario
  - Centre Hospitalier de l'Universite de Montreal (CHUM), Montreal, Quebec
  - CHA Hopital de I enfant-Jesus, Québec, Quebec
- China (26):
  - Beijing Cancer Hospital, Beijing
  - Peking University Third Hospital, Beijing
  - The First Hospital of Jilin University, Changchun
  - Hunan Cancer Hospital, Changsha
  - West China Hospital, Sichuan University, Chengdu
  - Sichuan Provincial People's Hospital, Chengdu
  - Second Affiliated Hospital of Third Military Medical University, Chongqing
  - Fujian Cancer Hospital, Fuzhou
  - Southern Medical University Nanfang Hospital, Guangdong Province Guangzhou City
  - Sun yat-sen University Cancer Center, Guangzhou
  - Zhujiang Hospital, Southern Medical University, Guangzhou
  - Harbin Medical University Cancer Hospital, Harbin
  - Anhui Province Cancer Hospital, Hefei
  - Shandong Cancer Hospital, Jinan
  - Jiangxi Cancer Hospital, Nanchang
  - Guangxi Cancer Hospital of Guangxi Medical University, Nanning
  - Fudan University Shanghai Cancer Center, Shanghai
  - First Hospital of China Medical University, Shenyang
  - Shengjing Hospital of China Medical University, Shenyang
  - First Affiliated Hospital of Soochow University, Suzhou
  - Institute of Hematology and Blood Diseases Hospital Chinese Academy of Medical Sciences, Tianjin
  - Tianjin Cancer Hospital, Tianjin
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan
  - Tongji Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan
  - The First Affiliated Hospital of Xiamen University, Xiamen
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou
- Denmark (3):
  - Aalborg Universitetshospital, Aalborg
  - Aarhus Universitetshospital Skejby, Aarhus N
  - Regionshospitalet Gødstrup, Herning
- France (10):
  - CHRU de Lille - Hopital Claude Huriez, Lille
  - Hospices Civils de Lyon, Lyon
  - Institut Paoli Calmettes, Marseille
  - CHU Montpellier, Montpellier
  - CHU de Nantes - Hotel Dieu, Nantes
  - CHU de Bordeaux, Pessac
  - CHU DE RENNES - CHU Pontchaillou, Rennes
  - Centre Henri Becquerel, Rouen
  - CHU Strasbourg Hpital Hautepierre, Strasbourg
  - IUCT Oncopole, Toulouse
- Germany (17):
  - Charité Universitätsmedizin Berlin, Berlin
  - Staedisches Klinikum Brandenburg, Brandenburg
  - Klinikum Chemnitz gGmbH, Klinik f. Innere Medizin III, Chemnitz
  - Universitätsklinikum Köln, Cologne
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Universitätsklinikum Erlangen, Medizinische Klinik 5, Hämatologie und Internistische Onkologie, Erlangen
  - Universitätsklinikum Essen, Essen
  - Universitätsklinikum Frankfurt, Frankfurt
  - UKE Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Universitaetsklinikum Schleswig Holstein - Campus Luebeck, Lübeck
  - Otto von Guericke Uni Magdeburg Uniklinik, Magdeburg
  - Klinikum rechts der Isar der TU München, III. Medizinische Klinik, München
  - Universitätsklinikum Münster, Münster
  - Klinikum Ernst von Bergman, Potsdam
  - Klinikum Stuttgart Katharinenhospital, Stuttgart
  - Universitätsklinikum Ulm, Ulm
  - Universitätsklinikum Würzburg, Würzburg
- Italy (9):
  - Istituto Nazionale Tumori Irccs Fondazione g. Pascale, Napoli, Campania
  - Policlinico S.Orsola-Malpighi, Bologna, Emilia-Romagna
  - A.O. Universitaria Policlinico Di Modena, Modena, Emilia-Romagna
  - A.O. Universitaria S. Martino Di Genova, Genoa, Liguria
  - Asst Papa Giovanni Xxiii, Bergamo, Lombardy
  - Fond. IRCCS Istituto Nazionale Tumori, Milan, Lombardy
  - Istituto Clinico Humanitas, Rozzano, Lombardy
  - A. O. U. Policlinico G. Rodolico, Catania, Sicily
  - Ospedale San Bortolo, Vicenza, Veneto
- Japan (24):
  - Anjo Kosei Hospital, Aichi
  - Aichi Cancer Center, Aichi
  - Nagoya University Hospital, Aichi
  - Chiba Cancer Center, Chiba
  - National Cancer Center Hospital East, Chiba
  - National Hospital Organization Kyushu Cancer Center, Fukuoka
  - Kyushu University Hospital, Fukuoka
  - Gifu University Hospital, Gifu
  - Hokkaido University Hospital, Hokkaido
  - Kobe City Medical Center General Hospital, Hyōgo
  - Kanagawa Cancer Center, Kanagawa
  - Tokai University Hospital, Kanagawa
  - University Hospital Kyoto Prefectural University of Medicine, Kyoto
  - Tohoku University Hospital, Miyagi
  - Okayama University Hospital, Okayama
  - Osaka Metropolitan University Hospital, Osaka
  - Kansai Medical University Hospital, Osaka
  - Kindai University Hospital, Osaka
  - Shimane University Hospital, Shimane
  - National Cancer Center Hospital, Tokyo
  - Komagome Hospital, Tokyo
  - The Cancer Institute Hospital of JFCR, Tokyo
  - Keio University Hospital, Tokyo
  - Yamagata University Hospital, Yamagata
- Mexico (4):
  - Health Pharma Professional Research, Mexico City, Mexico CITY (federal District)
  - Inst. Nacional de Cancerologia, Mexico City, Mexico CITY (federal District)
  - Hospital General de Mexico, Mexico, Tlaxcala
  - Hospital de Especialidades Centro Medico Nacional La Raza, Mexico City
- Poland (6):
  - Szpital Specjalistyczny Podkarpacki O?rodek Onkologiczny, Brzozów
  - Uniwersyteckie Centrum Kliniczne, Gda?sk
  - Pratia Onkologia Katowice, Katowice
  - ?wi?tokrzyskie Centrum Onkologii SPZOZ, Kielce
  - PRATIA MCM Kraków, Krakow
  - Uniwersytecki Szpital Kliniczny im. Jana Mikulicza-Radeckiego we Wroclawiu, Wroc?aw
- Auxilio Mutuo Cancer Center, San Juan, Puerto Rico
- South Korea (13):
  - Inje university Haeundae Paik Hospital, Busan
  - Pusan National University Hospital, Busan
  - Keimyung University Dongsan Medical Center, Daegu
  - Chungnam National University Hospital, Daejeon
  - National Cancer Center, Goyang-si
  - Chonnam National University Hwasun Hospital, Jeollanam-do
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Seoul St Mary's Hospital, Seoul
  - Yeouido St. Mary's Hospital, Seoul
- Spain (8):
  - Complejo Hospitalario Universitario de Santiago (CHUS), Santiago de Compostela, LA Coruna
  - Hospital Quiron de Madrid, Pozuelo de Alarcón, Madrid
  - Clinica Universitaria de Navarra, Pamplona, Navarre
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Clinica Universidad de Navarra Madrid, Madrid
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Clinico Universitario de Valencia, Valencia
- Universitaetsspital Basel, Basel, Switzerland
- Taiwan (6):
  - Chang Gung Medical Foundation - Chai Yi, Chai Yi
  - Chang Gung Medical Foundation - Kaohsiung;Oncology, Kaoisung
  - E-Da Cancer Hospital, Kaoshiung
  - China Medical University Hospital, Taichung
  - Chi-Mei Hospital, Liouying, Tainan
  - National Taiwan University Hospital, Taipei
- Turkey (Türkiye) (5):
  - Abdurrahman Yurtarslan Onkoloji Training and Research Hospital, Ankara
  - Ankara Universitesi Tip Fakultesi Hastaneleri - Cebeci Hastanesi, Ankara
  - Istanbul VKV American Hospital, Istanbul
  - Marmara University Pendik Training and Research Hospital, Istanbul
  - Kocaeli Univesity Medical Faculty, İzmit
- United Kingdom (11):
  - Barnet Hospital, Barnet
  - Blackpool Victoria Hospital, Blackpool
  - East Kent Hospitals University NHS Foundation Trust, Canterbury
  - Royal Devon and Exeter Hospital, Exeter
  - Beatson West of Scotland Cancer Centre, Glasgow
  - Leeds Teaching Hosp NHS Trust, Leeds
  - University College London Hospitals NHS Foundation Trust - University College Hospital, London
  - Guy'S Hospital, London
  - Newcastle University, Newcastle
  - Nottingham University Hospitals NHS Trust, Nottingham
  - Churchill Hospital - Oxford Cancer & Haematology Centre, Oxford

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing